CLINICAL TRIAL: NCT02053077
Title: A Study to Identify Risks in Routine Use of the GlucoTab System for Glycaemic Management in Non-critically Ill Patients With Type 2 Diabetes at General Wards
Brief Title: Risk Identification of the GlucoTab System in Routine Use
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, Univ. Prof. Dr., Medical University of Graz
Other Study IDs: ClinDiab-05
Record Dates: First submitted 2014-01-29; First posted 2014-02-03 (Estimated); Results first posted 2021-02-08 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Identification of risks of the GlucoTab system in routine use.

DETAILED DESCRIPTION:
A study to identify risks in routine use of the GlucoTab system for glycaemic management in non-critically ill patients with type 2 diabetes at general wards.

ELIGIBILITY:
Inclusion Criteria:

* informed consent obtained after being advised of the nature of the study
* type 2 diabetes or new-onset hyperglycaemia which require s.c. insulin therapy during hospital stay
* diabetes therapy supported by GlucoTab system

Exclusion Criteria:

* type 1 diabetes mellitus
* intravenous insulin therapy
* hyperglycaemic episodes (ketoacidosis, hyperosmolar state) if they require intravenous insulin therapy
* gestational diabetes or pregnancy
* known or suspected allergy to certain insulin types, named in the user manual
* total parenteral nutrition (TPN)
* any mental condition rendering the patient incapable of giving his consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-critically ill patients with type 2 diabetes at general wards
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2014-02; Primary Completion 2016-06 (Actual); Study Completion 2016-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R. Pieber, Univ.Prof.Dr, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Diabetes therapy was performed according to the intended use of the GlucoTab system
Period: Overall Study
Arm/Group | Intervention
Started | 150
Completed | 150
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56
  Male | 94

OUTCOME MEASURES:

1. Primary Outcome: Efficacy: Blood Glucose During Hospital Stay, an Expected Average of 1 Week
Description: efficacy: mean daily blood glucose during hospital stay, an expected average of 1 week
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 1 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intervention
Number analyzed (Participants) | 150
mg/dl | 159 (32)

2. Secondary Outcome: Efficacy: Blood Glucose During Hospital Stay
Description: Efficacy: mean pre-breakfast blood glucose during hospital stay
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 1 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Intervention
Number analyzed (Participants) | 150
mg/dl | 147 (38)

3. Secondary Outcome: Usability: Coverage of the GlucoTab
Description: Usability: coverage of the GlucoTab treatment during hospital stay
Time Frame: Participants will be followed for the duration of hospital stay, an expected average of 1 week
Population: Diabetes therapy was performed according to the intended use of the GlucoTab system
Measure: Mean (Standard Deviation); unit: percentage of hospital stay
Arm/Group | Intervention
Number analyzed (Participants) | 150
percentage of hospital stay | 71.4 (23.4)

ADVERSE EVENTS:
Time Frame: during hospital stay
Arm/Group | Intervention
Serious Adverse Events (participants affected / at risk) | 1/150
Other Adverse Events (participants affected / at risk) | 3/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=150)
Pneumonia and cardiac decompensation requiring treatment in intensive care unit (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=150)
Cystitis (Infections and infestations) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
AV Block Grad 3 (Cardiac disorders) | 1 (1)
Haemorrhagic Gastritis (Gastrointestinal disorders) | 1 (1)
Antibiotic associated exanthema (Skin and subcutaneous tissue disorders) | 1 (1)
Insult (Posteriorinfarction after intracardiac catheter) (Vascular disorders) | 1 (1)
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 1 (1)
Cholecystolithiasis (Hepatobiliary disorders) | 1 (1)
Aneurysma spurium right groin (Vascular disorders) | 1 (1)
NSTEMI (Cardiac disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Spondylodicscitis LWS (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes